CLINICAL TRIAL: NCT01761708
Title: Case-control Study of Mesh-infection After a Size Tailored Hernia Repair With C-Qur V-Patch
Acronym: Re-SITUP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Stijn De Sutter, Dr. Stijn De Sutter, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: Re-situp
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Ventral Hernia; Umbilical Hernia; Epigastric Hernia; Trocar-site Hernia
Keywords: primary ventral hernia repair with mesh; umbilical hernia repair; epigastric hernia repair; C-Qur V-patch; Size tailored repair; preperitoneal repair; abdominal hernia; dual sided mesh; trocar-site hernia
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical; Hernia, Abdominal | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- umbilical, epigastric and trocar-site hernia
  Interventions: Procedure: primary ventral hernia repair with mesh

INTERVENTIONS:
Procedure: primary ventral hernia repair with mesh

SUMMARY:
Ventral hernias, such as umbilical, epigastric and trocar-site hernias, are best repaired with abdominal wall reinforcement by mesh implantation. Mesh-devices using a dual-sided mesh technology have been developed for the specific indication of small ventral hernias; this technique is very attractive because the mesh can be introduced through a nearly invisible scar in the umbilicus. The dual layer of the mesh inhibits the formation of adhesions of the viscera to the mesh so, if wanted, it can be positioned in a intraperitoneal position. No literature is available on the adequate size of mesh needed to repair a hernia defect of an umbilical or epigastric hernia. Very small hernias are now often enlarged for repair with a large mesh device. Small hernias might benefit of repair with a small mesh device so no enlargement of the defect is necessary Larger hernias might benefit from a larger mesh size to have more overlap of the mesh beyond the hernia defect. The SITUP-trial was a prospective cohort study who was designed to explore the efficacy of C-QUR V-Patch of different sizes for the different sizes of hernia defects. The study was stopped prematurely because of the perception of an unacceptably high rate of mesh infection. This new study will retrospectively examine the incidence of mesh infection in all ventral hernias repaired with a C-QUR V-Patch. Collection of patient data was done using the Eura-HS registry.

ELIGIBILITY:
Inclusion Criteria:

all adult patients that are planned for surgical repair of a umbilical, epigastric or trocar-site hernia will be considered to enter the study.

Exclusion Criteria:

patients refusing to participate at the follow up visits pregnancy age < 18 years life expectancy less than 12 months emergency operations liver cirrhosis or ascites cancer patients concomitant surgery other than hernia repair

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
mesh infection | incidence over 12 months

SECONDARY OUTCOMES:
hernia recurrence rate | incidence over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stijn De Sutter, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares; Filip Muysoms, MD, Study Director — Algemeen Ziekenhuis Maria Middelares; Iris Kyle-Leinhase, PhD, Study Chair — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium